CLINICAL TRIAL: NCT04396093
Title: Analysis of Anxiety-depressive Patterns, Quality of Life and Personality Assessment in Patients With Pancreatic Cancer: Outcome of Adaptation to Disease and Clinical Treatments
Brief Title: Analysis Of The Anxiety-Depressive Pattern, Quality Of Life And Assessment Of Personality in Patients With Pancreatic Ductal Adenocarcinoma (PACT24)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Michele Reni (Other)
Responsible Party: Sponsor-Investigator, Michele Reni, MD, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: PACT24
Record Dates: First submitted 2020-05-13; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Pancreas Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: psychological support — specific questionnaires administration: EORTC QLQ 30, EORTC- PAN 26, HADS, Millon Clinical Multiaxial Inventory

SUMMARY:
The aim of this study is the evaluation of psychological aspects, such as anxiety-depressive patterns, quality of life, personality and other psychopathological syndromes of patients who receive a diagnosis of pancreatic cancer and who face chemotherapy treatment, radio-chemotherapy or surgery

DETAILED DESCRIPTION:
Pancreatic cancer is an aggressive disease whose prognosis is generally unfavorable: less than 20% of patients results eligible for resection treatment with potentially curative purposes and only in 2019 in Italy 13,500 new cases were estimated. It represents one of the poorest prognosis with 8.1% survival at 5 years and 3% at 10 years.

Its treatments can have a negative effect on the quality of life linked to the health of patients (HRQoL). Over the past 20 years, the quality of life assessment has become an important component of evaluating new therapeutic approaches, providing indications on the patient's perception of the benefits of the treatments to which he undergoes. Therefore, an accurate assessment of HRQoL using valid and standardized tools is crucial to highlight the costs and benefits of the different therapeutic options and the clinical utility of the data.

Description of the intervention (schedule of visits):

Visit 1 (screening). Patients will be informed about the study. Once patients agree with the inclusion in the study the investigators will evaluate the inclusion and exclusion criteria. Those patients who meet all the inclusion criteria and none of the exclusion criteria will be finally included in the study. In this visit, patients, tumor-related variables, and general patients' features will be recorded, and all questionnaires will be administered EORTC QLQ 30, EORTC- PAN 26, HADS, Millon Clinical Multiaxial Inventory).

Enrolled patients will make a first psychological visit within one month of the initial diagnosis and before starting active medical treatment (chemotherapy, radiochemotherapy, surgery). During this visit, they will be asked to complete questionnaires aimed at assessing the quality of life (EORCT QLQ 30, EORCT PAN26) of the anxiety-depressant aspects related to the disease (HADS) and of the personological functioning (MCMI-III) to proceed psychological evaluation.

During the visit 2 (2-3 months after the first dose of planned chemotherapy and following an instrumental re-evaluation), the quality of life and the anxiety-depression symptoms related to the disease will be re-evaluated (EORCT QLQ 30, EORCT PAN26; HADS)

The researcher will record in a dedicated database all patient information, such as:

* Personal data (gender, age, schooling)
* Onset and related timing of anxiety disorders or mood before the disease onset
* Psychological or psychiatric visits before the disease onset
* Psychotropic drugs use/abuse
* Psychotherapeutic or psychological path in progress
* Family, social, religious /spiritual resources
* Eligibility for surgery
* Stage of illness
* Clinical treatment (type of chemotherapy, radiochemotherapy)
* Therapeutic result (response, progression stability)
* Any serious adverse events (SAE).

The same variables recorded at Visit 1 will be checked again.

Power size calculation:

The number of patients was calculated taking into account the main outcome. Assuming a positive correlation coefficient of 0.3 (effect size) between the change in anxiety depression levels and self-perceived quality of life, an 85% power, a 5% significance level and a drop-out percentage / missing data equal to 30%, it is estimated a sample size of 75 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients candidated to receive an active treatment (surgery, chemiotherapy, chemio-radiation)
* Patients able to sign the informed consent.

Exclusion Criteria:

* • Patients with a school education level less than 8 years, since the complexity of submitted questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a confirmed diagnosis of pancreatic ductal adenocarcinoma (resectable, borderline resectable, locally advanced or metastatic)
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-05-10 (Estimated); Study Completion 2021-05-10 (Estimated)

PRIMARY OUTCOMES:
Analysis of the anxiety and depression in patients who face active cancer treatment (chemotherapy, radiotherapy, surgery) | 12 weeks after the diagnosis
  The prevalence and variations of the anxious and depressive symptoms related to the disease condition (HADS questionnaire) during the disease course
Analysis of the quality of life in patients who face active cancer treatment (chemotherapy, radiotherapy, surgery) | 12 weeks after the diagnosis
  The quality of life self-perceived by the patient (EORTC QLQ 30 - PAN 26 questionnaires) and its variations during the disease path

SECONDARY OUTCOMES:
The influence of patient personality on chemioterapic treatment response | 12 weeks after the diagnosis
  The influence of a maladaptive personality profiles and psychopathological aspects vs adaptive personality profiles and absence of disease psychopathological aspects (Millon Cutt off <75) on the quality of self-perceived life (EORTC QLQ 30 questionnaire) and on disease-related anxiety-depressive symptoms (HADS questionnaire) during the treatment through a psychodiagnostic assessment

CONTACTS AND LOCATIONS:
Overall Officials: Michele Reni, MD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS S Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Angelino AF, Treisman GJ. Major depression and demoralization in cancer patients: diagnostic and treatment considerations. Support Care Cancer. 2001 Jul;9(5):344-9. doi: 10.1007/s005200000195. PMID 11497387
- [Background] Brunault P, Champagne AL, Huguet G, Suzanne I, Senon JL, Body G, Rusch E, Magnin G, Voyer M, Reveillere C, Camus V. Major depressive disorder, personality disorders, and coping strategies are independent risk factors for lower quality of life in non-metastatic breast cancer patients. Psychooncology. 2016 May;25(5):513-20. doi: 10.1002/pon.3947. Epub 2015 Sep 10. PMID 26356037
- [Background] Champagne AL, Brunault P, Huguet G, Suzanne I, Senon JL, Body G, Rusch E, Magnin G, Voyer M, Reveillere C, Camus V. Personality disorders, but not cancer severity or treatment type, are risk factors for later generalised anxiety disorder and major depressive disorder in non metastatic breast cancer patients. Psychiatry Res. 2016 Feb 28;236:64-70. doi: 10.1016/j.psychres.2015.12.032. Epub 2015 Dec 25. PMID 26747215
- [Background] Fitzsimmons D, Johnson CD, George S, Payne S, Sandberg AA, Bassi C, Beger HG, Birk D, Buchler MW, Dervenis C, Fernandez Cruz L, Friess H, Grahm AL, Jeekel J, Laugier R, Meyer D, Singer MW, Tihanyi T. Development of a disease specific quality of life (QoL) questionnaire module to supplement the EORTC core cancer QoL questionnaire, the QLQ-C30 in patients with pancreatic cancer. EORTC Study Group on Quality of Life. Eur J Cancer. 1999 Jun;35(6):939-41. doi: 10.1016/s0959-8049(99)00047-7. PMID 10533475
- [Background] Fras I, Litin EM, Bartholomew LG. Mental symptoms as an aid in the early diagnosis of carcinoma of the pancreas. Gastroenterology. 1968 Aug;55(2):191-8. No abstract available. PMID 4385690
- [Background] Green AI, Austin CP. Psychopathology of pancreatic cancer. A psychobiologic probe. Psychosomatics. 1993 May-Jun;34(3):208-21. doi: 10.1016/S0033-3182(93)71882-4. PMID 8493302
- [Background] Gupta D, Lis CG, Grutsch JF. The European organization for research and treatment of cancer quality of life questionnaire: implications for prognosis in pancreatic cancer. Int J Gastrointest Cancer. 2006;37(2-3):65-73. doi: 10.1007/s12029-007-0001-9. PMID 17827524
- [Background] Kelsen DP, Portenoy RK, Thaler HT, Niedzwiecki D, Passik SD, Tao Y, Banks W, Brennan MF, Foley KM. Pain and depression in patients with newly diagnosed pancreas cancer. J Clin Oncol. 1995 Mar;13(3):748-55. doi: 10.1200/JCO.1995.13.3.748. PMID 7884435
- [Background] Passik SD, Roth AJ. Anxiety symptoms and panic attacks preceding pancreatic cancer diagnosis. Psychooncology. 1999 May-Jun;8(3):268-72. doi: 10.1002/(SICI)1099-1611(199905/06)8:33.0.CO;2-W. PMID 10390740